CLINICAL TRIAL: NCT04917341
Title: The Compatibility of Preoperative Endometrial Biopsies With Postoperative Final Pathology in Endometrial Cancer; Should Preoperative Pathology Samples of Patients Referred to a Tertiary Center be Re-evaluated?
Brief Title: The Compatibility of Preoperative Endometrial Biopsies With Postoperative Final Pathology in Endometrial Cancer
Status: Completed | Type: Observational
Sponsor: Batman Training and Research Hospital (Other Government)
Collaborators: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Erhan Okuyan,M.D, M.D, Batman Training and Research Hospital
Other Study IDs: 2020-12
Record Dates: First submitted 2021-05-27; First posted 2021-06-08 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Endometrial Cancer Stage; Gynecologic Cancer
Keywords: preoperative endometrial biopsies; postoperative final pathology; Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- preoperative endometrial sampling result (secondary hospital)/1: Endometrial biopsy samples taken at the stage 2 state hospital
  Interventions: Diagnostic Test: re-evaluation of endometrial biopsy samples by a gynecopathologist working at a university hospital
- preoperative endometrial sampling result (tertiary hospital)/2: Endometrial biopsy samples taken at the stage (tertiary hospital)
  Interventions: Diagnostic Test: re-evaluation of endometrial biopsy samples by a gynecopathologist working at a university hospital
- final postoperative pathology/3: final postoperative pathology results with grade (endometrium cancer)
  Interventions: Diagnostic Test: re-evaluation of endometrial biopsy samples by a gynecopathologist working at a university hospital

INTERVENTIONS:
Diagnostic Test: re-evaluation of endometrial biopsy samples by a gynecopathologist working at a university hospital — The endometrial biopsy samples taken at the second stage state hospital were re-evaluated by the gynecopathologist working at the university hospital and / or the repeated endometrial biopsy sampling was examined and the evaluation process was carried out in two steps.

SUMMARY:
Although there are many studies comparing preoperative and postoperative histological diagnoses in the literature, there are no studies evaluating the compatibility of preoperative histological diagnoses obtained from different centers with postoperative histological diagnoses.Therefore, in our study, we aimed to determine whether preoperative pathological specimens need to be re-evaluated in the referenced hospitals by comparing the compatibility of endometrial specimens in secondary care and tertiary centers with their final pathologies.In our study, we aimed to reveal the under and overdiagnosis rates of the preoperative histological diagnoses of our hospitals compared to the final pathology.

DETAILED DESCRIPTION:
Medical data of 960 patients diagnosed with endometrial cancer by endometrial biopsy between 2002 and 2016 were retrospectively analyzed. Of these patients, 41 were excluded from the study due to non-surgical treatment, 254 patients having biopsy only in one center preoperatively, and lack of medical data in 52 patients.The study included 613 patients who had preoperative endometrial biopsy specimens evaluated by two different centers, diagnosed with endometrial cancer and treated surgically. Our study was conducted in the gynecological oncology department of our university after obtaining the approval of the ethics committee numbered 430-2019.The clinicopathological characteristics of the patients were evaluated by examining the hospital records of age, gravida, parity, BM (body mass index), menopausal status and systemic diseases. Histopathological and clinical features of endometrial cancer were reviewed.In this study, endometrial biopsy samples taken in the second stage state hospital were re-evaluated by the gynecopathologist working at the university hospital and / or the evaluation process was carried out in two steps by examining the repeated endometrial biopsy sampling.Patients diagnosed with endometrial cancer were treated surgically in our clinic. Endometrial sampling results based on uterine cancer risk groups; While histologically endometrioid and nonendometrioid were evaluated in two groups, the greade1-2 (low risk), greade3 (high risk) of uterine cancer were evaluated in four groups as those without malingnancy (benign and premaling lesions).By comparing these preoperative histological diagnoses with postoperative surgical final pathology, the accuracy rates for histological type and greade were determined. In addition, lower diagnosis, comorbidity and higher diagnosis rates compared to final pathology were examined for two different centers.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 40-90 years diagnosed with endometrial cancer according to

endometrial sampling results

Exclusion Criteria:

* Lack of medical data
* Endometrial sampling in only one center

Ages: 40 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients aged 40-90 years diagnosed with endometrial cancer according to endometrial sampling results
Study Population: Patients who received treatment in a tertiary care center for cancer of endometry
Sampling Method: Probability Sample
Enrollment: 960 (Actual)
Dates: Start 2002-04-12 (Actual); Primary Completion 2021-04-24 (Actual); Study Completion 2021-05-27 (Actual)

PRIMARY OUTCOMES:
Comparison of endometrial sampling results performed in 2 different centers | 1 year
  in our study, we aimed to determine whether preoperative pathological specimens need to be re-evaluated in the referenced hospitals by comparing the compatibility of endometrial specimens in secondary care and tertiary centers with their final pathologies.

SECONDARY OUTCOMES:
To reveal the rates of under and overdiagnosis of preoperative histological results | 1 year
  Correlation of preoperative pathological diagnoses with postoperative final pathological diagnoses.

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf Cakmak, M.D, Principal Investigator — Batman education and research hospital

IPD SHARING:
Plan to Share IPD: No